CLINICAL TRIAL: NCT07287657
Title: Exploring the Impact of Transcutaneous Electrical Acupoint Stimulation Therapy on Postoperative Pain, Quality of Life, and Blood Inflammatory Markers in Lung Cancer Patients After Video Assisted Thoracoscopic Surgery
Brief Title: Exploring the Effects of Transcutaneous Electrical Acupoint Stimulation Therapy on Patients After Video-Assisted Thoracoscopic Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Lin,Chun-Ya
Record Dates: First submitted 2025-04-28; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative
Keywords: Video-assisted thoracoscopic surgery(VATS); Enhanced Recovery After Surgery(ERAS); pain, postoperative; transcutaneous electrical acupoint stimulation; transcutaneous electrical nerve stimulation; acute pain; blood inflammatory biomarkers; quality of life; Anxiety and Depression
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Anxiety Disorders; Depression | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Participants receive standard postoperative analgesia according to institutional protocol.
  Interventions: Drug: Standard Analgesia
- TENS Group (Experimental): Participants receive standard postoperative analgesia combined with transcutaneous electrical nerve stimulation (TENS)
  Interventions: Drug: Standard Analgesia; Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- TENS + TEAS Group (Experimental): Participants receive standard postoperative analgesia combined with both transcutaneous electrical nerve stimulation (TENS) and transcutaneous electrical acupoint stimulation (TEAS).
  Interventions: Drug: Standard Analgesia; Device: Transcutaneous Electrical Nerve Stimulation (TENS); Device: Transcutaneous Electrical Acupoint Stimulation (TEAS)

INTERVENTIONS:
Drug: Standard Analgesia — Postoperative analgesic medications administered according to standard clinical practice and hospital guidelines
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Non-invasive electrical nerve stimulation therapy applied to specific areas to reduce postoperative pain
  Arms: TENS + TEAS Group; TENS Group
Device: Transcutaneous Electrical Acupoint Stimulation (TEAS) — Electrical stimulation applied to specific acupuncture points through the skin to enhance analgesic efficacy and modulate autonomic function.
  Arms: TENS + TEAS Group

SUMMARY:
Thoracic surgery is known to be one of the most painful types of surgery. If acute postoperative pain is not properly managed, there is a high risk that it may develop into clinically significant chronic pain within six months after surgery, which can seriously affect quality of life. According to research on Enhanced Recovery After Surgery (ERAS), using multimodal pain management strategies can significantly reduce postoperative pain and decrease reliance on pain medications. This study aims to investigate whether combining transcutaneous Electrical Nerve Stimulation therapy with conventional pain management can further enhance pain relief and improve recovery outcomes.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of three postoperative analgesic strategies in patients undergoing lesion resection via video-assisted thoracoscopic surgery (VATS). Under standard postoperative care protocols, patients will be randomized into three groups: (1) conventional pharmacologic analgesia alone, (2) conventional analgesia combined with transcutaneous electrical nerve stimulation (TENS), and (3) conventional analgesia combined with both transcutaneous electrical nerve stimulation (TENS) and transcutaneous electrical acupoint stimulation (TEAS). The primary outcomes include the assessment of acute postoperative pain intensity, blood inflammatory biomarkers, health-related quality of life, and the incidence of postoperative complications. This investigation seeks to determine whether adjunctive use of neuromodulatory techniques such as TENS and TEAS can enhance analgesic efficacy and improve postoperative recovery profiles.

ELIGIBILITY:
Inclusion Criteria:

* People who are about to undergo thoracic surgery

Exclusion Criteria:

* Patients with epilepsy,
* Pacemaker installed
* Severe infections status

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity Assessed Using the Visual Analog Scale (VAS) | Within 48 hours after surgery
  Pain intensity will be assessed using a 10-point Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain."

SECONDARY OUTCOMES:
Blood Inflammatory Markers | Within 48 hours after surgery
  Blood inflammatory markers, including the neutrophil-to-lymphocyte ratio (NLR) and lymphocyte-to-monocyte ratio (LMR), will be calculated using complete blood count (CBC) parameters. NLR increases are commonly interpreted as indicators of elevated systemic inflammation, whereas decreases in LMR may reflect enhanced inflammatory activity or physiological stress following surgery. These ratios will be assessed at multiple perioperative time points to evaluate changes in inflammatory response. The relationship between postoperative pain levels, clinical recovery, and changes in NLR and LMR will be analyzed to determine whether inflammatory activation is associated with greater postoperative pain or adverse outcomes. Units of measure are expressed as ratios (NLR, LMR).
Hospital Anxiety and Depression Scale | At baseline (preoperative), and after surgery 6 and 48 hours later
  The Hospital Anxiety and Depression Scale (HADS) will be used to evaluate participants' psychological status during the perioperative period. The scale consists of 14 items, with 7 items assessing anxiety (HADS-A) and 7 items assessing depression (HADS-D). Each item is scored from 0 to 3, yielding subscale scores ranging from 0 to 21. Higher scores indicate greater levels of anxiety or depression. Changes in HADS-A and HADS-D scores will be analyzed to determine postoperative psychological responses and the potential impact of different analgesic interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Taipei, Hualien, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Because it is still underway, I will share it after the research is completed.

REFERENCES:
- [Background] Edwards DA, Hedrick TL, Jayaram J, Argoff C, Gulur P, Holubar SD, Gan TJ, Mythen MG, Miller TE, Shaw AD, Thacker JKM, McEvoy MD; POQI-4 Working Group. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Perioperative Management of Patients on Preoperative Opioid Therapy. Anesth Analg. 2019 Aug;129(2):553-566. doi: 10.1213/ANE.0000000000004018. PMID 30768461

DOCUMENTS (3):
  • Study Protocol (2025-12-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT07287657/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT07287657/SAP_001.pdf
  • Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT07287657/ICF_002.pdf